CLINICAL TRIAL: NCT05152238
Title: Multicenter National ITP Registry and Accompanying Biospecimen Collection
Brief Title: ITP Registry and Accompanying Biospecimen Collection
Acronym: ITP-Registry
Status: Recruiting | Type: Observational
Sponsor: Jena University Hospital (Other)
Collaborators: University Hospital Dresden (Other); Novartis (Industry); Swedish Orphan Biovitrum (Industry); Grifols Biologicals, LLC (Industry); Amgen (Industry); argenx (Industry)
Responsible Party: Principal Investigator, Thomas Stauch, Principal Investigator, Jena University Hospital
Other Study IDs: ZKSJ0142
Record Dates: First submitted 2021-11-23; First posted 2021-12-09 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — 18 mL whole blood (peripheral venipuncture) and 9 ml bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective of this ITP registry is to collect clinical information, including biosampling, from consenting patients with a variety of ITPs at different points in the course of their disease.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is a rare hematologic disorder that can lead to a greater risk of bleeding or a prolonged bleeding time due to an autoimmune-mediated deficiency of platelets.

In recent years, new treatment options for patients with immune thrombocytopenia have emerged.

The results of published clinical studies on ITP can only be used for broad patient care to a limited extent, as they are designed for a patient population with clearly defined inclusion and exclusion criteria. Real world data collected from this registry will help to better understand the diagnosis and therapy of ITP patients in everyday treatment and to more effectively direct individual patients to optimal therapy, thus improving their outcomes.

By collecting biospecimens, this project will contribute new knowledge to the study of ITP through standardized, systematic, and high-quality collection and storage of patient samples and associated data.

The registry collects clinical data from patients diagnosed with ITP at defined points in the course of the disease. The Data collection includes a range of clinical measures, disease-related factors, treatment/treatment course and outcomes, complications during treatment and Qol, fatigue scoring and survival data (up to 5 years).

The data are collected prospectively. In addition, patients can be included retrospectively up to 12 months after the initial diagnosis if continuous documentation can be provided at the treatment centre. In both cases, a written declaration of consent is obligatory.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary Immune Thrombocytopenia (ITP)
* Age ≥18 years
* signed declaration of consent

Exclusion Criteria:

* diagnoses that cannot be reconciled with the diagnosis of ITP (esp. heparin-induced thrombocytopenia, pregnancy-associated thrombocytopenia, pseudothrombocytopenia)
* no informed consent possible (this covers patients who are unable to understand the nature and scope of participation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Immune thrombocytopenia (ITP) which is a rare hematologic disorder that can lead to a greater risk of bleeding or a prolonged bleeding time due to an autoimmune-mediated deficiency of platelets. There is a distinction between a primary form, in which no triggering cause is identifiable, and secondary forms, which may for example occur in the context of systemic autoimmune diseases or drug-induced.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
epidemiological data on ITP - Incidence | At enrollment
  Incidence: number of reported ITP, estimate incidence by zip code area
epidemiological data on ITP - Age | At enrollment
  Age (year of birth)
epidemiological data on ITP - Sex distribution | At enrollment
  Sex distribution: female, male
Description of the causes of ITP | At enrollment
  causes of ITP in primary/secondary form (medical induced, autoimmune disease, Lymphoma / malignancy, infection, upon vaccination, others)
ITP treatment type received | 5 years
  Medical therapies received
Remission | 5 years
  Remission Status

SECONDARY OUTCOMES:
Recording of clinical characteristics of affected patients - Disease stage | At enrollment, 6 months, annually up to 5 years
  bleeding severity WHO-CTCAE Grade 1-4
Recording of clinical characteristics of affected patients- platelet counts | At enrollment, 6 months, annually up to 5 years
  platelet counts in Gpt/l
Recording of clinical characteristics of affected patients -disease manifestation at diagnosis | At enrollment
  Localisation of bleeding and severity (WHO-CTCAE Grading)
Bleeding events | At enrollment, 6 months, annually up to 5 years
  Bleeding events (yes, no)
thromboembolic events | At enrollment, 6 months, annually up to 5 years
  thromboembolic events (no, Deep vein thrombosis, acute pulmonary artery embolism, other)
Quality of Life questionaire | At enrollment, 6 months, annually up to 5 years
  ILQI questionaire
fatigue assessment | At enrollment, 6 months, annually up to 5 years
  FACIT-F questionaire: subscale fatigue (only last 13 questions)
Laboratory parameters ANA | At enrollment, 6 months, annually up to 5 years
  ANA (negative/positive)
Laboratory parameters APL-Antibodies | At enrollment, 6 months, annually up to 5 years
  APL-Antibodies (negative/positive)
Laboratory parameters Lupus-Antibodies | At enrollment, 6 months, annually up to 5 years
  lupus-Antibodies (negative/positive)
Laboratory parameters platelet autoantibodies | At enrollment, 6 months, annually up to 5 years
  platelet autoantibodies (negative/positive)
Laboratory parameters helicobacter pylori | At enrollment, 6 months, annually up to 5 years
  helicobacter pylori (negative/positive)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Stauch, Dr. med., Study Director — Jena University Hospital; Karolin Trautmann-Grill, Dr. med., Study Director — Dresden Univeristy Hospital
Locations (64):
- Germany (64):
  - Universitätsklinikum Aachen AöR, Aachen
  - Klinikum Altenburger Land GmbH, Klinik für Innere Medizin/Hämatologie/Onkologie, Altenburg
  - MVZ am Klinikum Aschaffenburg, Aschaffenburg
  - MVZ IMD GmbH, IMD Gerinnungszentrum Hochtaunus, Bad Homburg
  - Onkologie/Hämatologie, Bad Liebenwerda
  - Charité Universitätsmedizin Berlin, Berlin
  - Praxis für Hämatologie und Onkologie Berlin-Mitte, Berlin
  - Vivantes Netzwerk für Gesundheit GmbH, Klinikum am Friedrichshain, Berlin
  - Onkologie am Segelfliegerdamm, Berlin
  - MVZ Hämatologikum GmbH, Biberach
  - Augusta-Kranken-Anstalt gGmbH, Bochum
  - Klinikum Chemnitz gGmbH, Chemnitz
  - MVZ Klinikum Coburg GmbH, Coburg
  - Klinikum Darmstadt, Darmstadt
  - ARGE e.V., Donauwörth
  - Onkozentrum Dresden/Freiberg, Dresden
  - Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Gemeinschaftspraxis Mohm & Prange-Krex, Dresden
  - Universitätsklinikum Dresden, Dresden
  - Krankenhaus Düren gGmbH, Düren
  - Onkologische Praxis Erfurt, Erfurt
  - Universitätsklinikum Erlangen, Erlangen
  - MVZ für Hämatologie und Onkologie Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Haemostas-Frankfurt, Frankfurt am Main
  - PIOH Studien und Management GbR, Frechen
  - Fachärztliche Gemeinschaftspraxis Panagiotou/Minaei, Garbsen
  - IOGP Gera MVZ GmbH, Gera
  - ALB FILS Kliniken, Klinik am Eichert, Göppingen
  - Universitätsklinik Greifswald, Greifswald
  - Katholisches Krankenhaus Hagen gGmbH, Hagen
  - Gemeinschaftspraxis, FA für Innere Medizin, Halle
  - MVZ III Onkologie der evidia MVZ Halle (Saale) GmbH, Halle
  - Onko-Kolleg GmbH & Co. KG, HOPA MVZ GmbH, Hamburg
  - Werlhof-Institut MVZ GmbH, Hanover
  - Onkologie am Raschplatz, Hanover
  - Dres. Kamal & Dorn GbR, Hanover
  - ODZ-Petersen GmbH, Heidenheim
  - St. Bernward Krankenhaus GmbH, Hildesheim
  - Klinikum Idar-Oberstein GmbH, Idar-Oberstein
  - University Hospital Jena, Jena
  - Klinikum Kassel GmbH, Kassel
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Gemeinschaftsklinikum Mittelrhein gGmbH, Ev. Stift St. Martin, Koblenz
  - Ambulantes Zentrum für Hämatologie, Onkologie und Gerinnung, Kronach
  - MVZ mbH, Onkologische Schwerpunktpraxis, Leer
  - Universitätsklinikum Leipzig, Leipzig
  - OnkoFor Leipzig GmbH, Leipzig
  - Universitätsklinikum Magdeburg, Klinik für Hämatologie, Onkologie und Zelltherapie, Magdeburg
  - Carl-von-Basedow Klinikum Merseburg, Merseburg
  - Gemeinschaftspraxis Hämato-Onkologie, München
  - Dietrich-Bonhoeffer-Klinikum Neubrandenburg, Neubrandenburg
  - MVZ Onko Medical GmbH Neustadt, Neustadt am Rübenberge
  - Pi.Tri.-Studien GmbH, Offenburg
  - Elblandkliniken Stiftung & Co. KG, Elblandklinikum Riesa, Riesa
  - Klinikum Südstadt Rostock, Rostock
  - Medcenter Nordsachsen, Schkeuditz
  - MVZ am Schlossgarten, Zero Praxen, Schwetzingen
  - Onkologiezentrum Soest/Iserlohn, Soest
  - Bundeswehrkrankenhaus Ulm, Ulm
  - Schwarzwald-Baar. Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen
  - Onkologisches Zentrum Wolfsburg-Helmstadt MVZ GmbH, Wolfsburg
  - Universitätsklinikum Würzburg, Würzburg
  - Praxis für Hämatologie und Internistische Onkologie, Zittau

IPD SHARING:
Plan to Share IPD: No
There is no validated data sharing procedure at the university hospital Jena. But of course it is planned to share the results with scientific community and publish the data in a scientific journal.